CLINICAL TRIAL: NCT04699032
Title: A Phase 1, Open-Label Evaluation of the Pharmacokinetics and Safety of a Single Dose of Apraglutide in Subjects With Normal and Impaired Renal Function.
Brief Title: Study of Pharmacokinetics and Safety of Apraglutide in Participants With Normal and Impaired Kidney Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA799-014
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Disease
Keywords: Renal Function; Renal Impairment; Kidney Function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — apraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Severe Renal Impairment (Experimental): eGFR (mL/min/1.73 m2): <30 not on hemodialysis
  Interventions: Drug: Apraglutide
- Normal Healthy Match (Experimental): eGFR (mL/min/1.73 m2): ≥90
  Interventions: Drug: Apraglutide
- Moderate Renal Impairment (Experimental): eGFR (mL/min/1.73 m2): ≥30 to 60
  Interventions: Drug: Apraglutide
- Mild Renal Impairment (Experimental): eGFR (mL/min/1.73 m2): ≥60 to 90
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Single dose of apraglutide 5 mg.

SUMMARY:
Study of pharmacokinetics and safety of apraglutide in participants with normal and impaired kidney function.

DETAILED DESCRIPTION:
A two stage design, open label, multi-center, non-randomized trial to evaluate the PK and safety of a single subcutaneous dose of 5 mg apraglutide in subjects with varying degrees of renal function. The renal function was calculated by the estimated glomerular filtration rate (eGFR) according to the Chronic Kidney Disease Epidemiology (CKD-EPI) Creatinine Equation.

Part 1: 8 subjects with severe renal impairment (Cohort 1) and 8 subjects with normal renal function (Cohort 2).

Part 2: 8 subjects with moderate (Cohort 3) and 8 subjects with mild (Cohort 4). Enrollment into Part 2 was conditional on the results of Part 1.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Age between 18 and 75 years inclusive
* Subjects who are willing and able to comply with the study procedures
* Subjects able to understand and willing to sign the informed consent
* Body mass index (BMI) of ≥17.5 to ≤40 kg/m2; and a total body weight of >50 kg (110 lb).
* Women of childbearing potential (WOCBP) on highly effective method of contraception during the trial and for 1 month after the end of trial (EOT) visit. Sterilized or infertile or postmenopausal females.
* Male subjects with a female partner of childbearing potential: highly effective methods of contraception and no sperm donation during the trial and for 1 month after (EOT) visit.

Healthy participants

* No clinically relevant abnormalities (medical history, vital signs, ECG, safety labs)
* eGFR measured by CKD-EPI ≥90 mL/min/1.73 m2) at two screening visits
* Demographically comparable to the group of subjects with impaired renal function:

Participants with impaired renal function

* Severe renal impairment: eGFR <30 mL/min/1.73 m2, but not requiring hemodialysis
* Moderate renal impairment: eGFR ≥30 mL/min/1.73 m2 and <60 mL/min/1.73 m2
* Mild renal impairment: eGFR ≥60 and <90 mL/min/1.73 m2

Exclusion Criteria:

All Subjects

* Renal transplant recipients
* History of systemic infection
* Any active malignancies or history of malignancies within the past 2 years
* Acute or chronic medical or psychiatric condition
* Treatment with an IMP within 30 days or 5 half-lives (whichever is longer) preceding the dose of IMP
* Male subjects partners of WOCBP who are unable to comply with the contraceptive measures
* History of clinically significant intestinal adhesions and/or chronic abdominal pain
* History of known colon polyps or family history of familial adenomatous polyposis
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen or human immunodeficiency virus (HIV)-1 and -2 antibodies
* Serum albumin concentration <25 g/L (2.5 g/dL)
* Hemoglobin concentration <90 g/L (9.0 g/dL)
* Aspartate amino transaminase (AST) or alanine amino transaminase (ALT) values >2 × upper limit of normal (ULN)
* Proteinuria of >3 g total bilirubin >1.5 × ULN
* Positive urine test for alcohol or illicit drugs at either Screening or admission.
* Clinically significant abnormalities on 12-lead ECG
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or five half-lives (whichever is longer) prior to Day 1. Stable concomitant medications may be given to subjects with renal impairment, if they are considered necessary for the welfare of the subjects.
* History of regular alcohol consumption exceeding seven drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine, or 12 ounces [360 mL] of beer, or 1.5 ounces [45 mL] of hard liquor) within 3 months of Screening
* Female subjects of childbearing potential who are unwilling or unable to use highly effective methods of contraception for the duration of the trial and for at least 1 month after the administration of the IMP; pregnant female subjects; female subjects planning to become pregnant during the duration of the trial and until 1 month after the administration of the IMP; breastfeeding female subjects
* Blood donation of approximately 500 mL or more within 60 days prior to the dose of IMP. Plasma donations of approximately 500 mL or more within 28 days prior to the dose of IMP

Additional Exclusion Criteria for Healthy Subjects with Normal Renal Function

* Evidence or history of clinically significant abnormalities
* Evidence or history of clinically significant dermatological condition

Additional Exclusion Criteria for Subjects with Impaired Renal Function

* Subjects requiring hemodialysis and/or peritoneal dialysis
* Subjects with other clinically significant disease
* Subjects with any significant hepatic, cardiac, or pulmonary disease or subjects who are clinically nephrotic. Hypertension, diabetes mellitus, hyperparathyroidism, ischemic heart disease are not cause for exclusion as long as the subject is medically stable and any drugs that are administered for these conditions are not expected to interfere with the PK of apraglutide.
* Screening BP ≥180 mmHg (systolic) or ≥110 mmHg (diastolic)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Clinical Research, Inc., Saint Paul, Minnesota

REFERENCES:
- [Derived] Greig G, Youssef NN, Bolognani F. Pharmacokinetics and Tolerability of a Single Dose of Apraglutide, a Novel, Long-Acting, Synthetic glucagon-like peptide-2 Analog With a Unique Pharmacologic Profile, in Individuals With Impaired Renal Function. J Clin Pharmacol. 2024 Jun;64(6):744-754. doi: 10.1002/jcph.2423. Epub 2024 Mar 11. PMID 38465515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed in the United States of America between 08 December 2020 and 05 July 2021.
Pre-assignment Details: 16 participants were included in Part 1 of the study and received 5 mg subcutaneous (SC) apraglutide on Day 1. Of the 16 participants who were included in Part 1, eight had normal renal function and eight had severely impaired renal function. Enrollment into Part 2 of the study was conditional on the results of Part 1. No participants were enrolled into Part 2.
Groups:
- Severely Impaired Renal Function: Participants with eGFR values <30 mL/min/1.73 m^2, but not requiring hemodialysis, received 5 mg SC apraglutide on Day 1.
- Normal Renal Function: Participants with estimated glomerular filtration rate (eGFR) values ≥90 mL/min/1.73 m^2 received 5 mg SC apraglutide on Day 1.
Period: Overall Study
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Normal Renal Function: Participants with eGFR values ≥90 mL/min/1.73 m^2 received 5 mg SC apraglutide on Day 1.
- Total: Total of all reporting groups
Arm/Group | Severely Impaired Renal Function | Normal Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] | 66 [54 to 75] | 60 [56 to 70] | 63 [54 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Full Range); unit: kg] | 90.1 [77.7 to 98.2] | 86.7 [76.2 to 98.4] | 88.4 [76.2 to 98.4]
Height [Mean (Full Range); unit: cm] | 171.9 [164.5 to 178.5] | 174.9 [168.5 to 181.0] | 173.4 [164.5 to 181.0]
Body mass index [Mean (Full Range); unit: kg/m^2] | 30.6 [24.4 to 33.7] | 28.3 [25.8 to 31.5] | 29.4 [24.4 to 33.7]
Estimated glomerular filtration rate [Mean (Full Range); unit: mL/min/1.73m^2] | 21.3 [11.4 to 28.5] | 96.3 [91.4 to 108.0] | 58.8 [11.4 to 108.0]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Apraglutide
Description: Pharmacokinetic (PK) samples collected for the measurement of plasma concentration of apraglutide were analyzed using a validated analytical method in compliance with applicable standard operating procedures.
Time Frame: 5 minutes pre-dose up to 240 hours after dosing on Day 1
Population: The PK parameter analysis population included all participants assigned to the investigational medicinal product (IMP) who were treated and had at least one of the PK parameters of primary interest measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
Number analyzed (Participants) | 8 | 8
ng/mL | 39.5 (13.7) | 65.8 (37.5)
Statistical Analysis 1: Comparison: Severely Impaired Renal Function vs Normal Renal Function; Test type: Other — Analysis of variance (ANOVA) was used to compare the natural log transformed Cmax for apraglutide between normal renal function group (Reference) and the severe impaired renal group (Test). Estimates of the mean differences and corresponding 90% confidence intervals (CIs) were obtained from the model. The mean differences and 90% CIs for the mean differences were exponentiated to provide estimates of the geometric least-square mean ratio (Test/Reference) and 90% CIs for the ratios; Geometric least-square mean ratio = 0.620, 90% CI 2-sided [0.423 to 0.909]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of Apraglutide
Description: PK samples collected for the measurement of plasma concentration of apraglutide were analyzed using a validated analytical method in compliance with applicable standard operating procedures.
Time Frame: 5 minutes pre-dose up to 240 hours after dosing on Day 1
Population: The PK parameter analysis population included all participants assigned to the IMP who were treated and had at least one of the PK parameters of primary interest measured.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL | 3330 (1150) | 5050 (3170)
Statistical Analysis 1: Comparison: Severely Impaired Renal Function vs Normal Renal Function; Test type: Other — ANOVA was used to compare the natural log transformed AUCinf for apraglutide between normal renal function group (Reference) and the severe impaired renal group (Test). Estimates of the mean differences and corresponding 90% CIs were obtained from the model. The mean differences and 90% CIs for the mean differences were exponentiated to provide estimates of the geometric least-square mean ratio (Test/Reference) and 90% CIs for the ratios; Geometric least-square mean ratio = 0.694, 90% CI 2-sided [0.458 to 1.050]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) that occurred after dosing the participant with the study drug. Participants with more than one TEAE were counted only once using the most severe event. Vital signs, triplicate 12-lead electrocardiograms, or clinical laboratory assessments considered clinically significant by the Investigator were reported as AEs.
Time Frame: Day 1 up to Day 14
Population: The Safety Set included all participants who received at least one dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants | 3 | 2

4. Secondary Outcome: Number of TEAEs
Description: The Investigator used the adjectives mild, moderate, or severe to describe the maximum intensity of the AE. These were defined as follows:
  * Mild: did not interfere with participant's usual function
  * Moderate: interfered to some extent with participant's usual function
  * Severe: interfered significantly with participant's usual function.
  The Investigator systematically assessed the causal relationship of AEs to IMP/trial treatment using the definitions below:
  * Not related: Not reasonably related to the IMP. The AE could not medically (pharmacologically/clinically) be attributed to the IMP
  * Related: Reasonably related to the IMP. The AE could medically (pharmacologically/clinically) be attributed to the IMP.
  A serious AE (SAE) was classified as any AE that:
  * Resulted in death
  * Was life-threatening
  * Required or prolonged in-patient hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect in a neo
Time Frame: Day 1 up to Day 14
Population: The Safety Set included all participants who received at least one dose of the IMP.
Measure: Number; unit: events
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
Number analyzed (Participants) | 8 | 8
events
  Any TEAEs | 7 | 3
  Any Mild TEAEs | 4 | 1
  Any Moderate TEAEs | 3 | 2
  Any Severe TEAEs | 0 | 0
  Any Treatment-Related TEAEs | 5 | 0
  Any Serious TEAEs | 0 | 0
  Any TEAEs leading to study discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 14
Description: The Safety Set included all participants who received at least one dose of the IMP.
Arm/Group | Severely Impaired Renal Function | Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severely Impaired Renal Function (N=8) | Normal Renal Function (N=8)
Chest pain (General disorders) | 1 (1) | 0 (0)
Injection site hemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site papule (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT04699032/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04699032/SAP_001.pdf